CLINICAL TRIAL: NCT05621564
Title: The Effect of Pre-operative Therapy on Response and Survival in Breast Cancer
Brief Title: Pre-operative Therapy in Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Wenjin Yin, Deputy Chief of Breast Surgery Department, RenJi Hospital
Other Study IDs: LY2022-028-B
Record Dates: First submitted 2022-11-08; First posted 2022-11-18 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- early breast cancer: no requirements for therapy
  Interventions: Drug: pre-operative therapy
- advanced breast cancer: no requirements for therapy
  Interventions: Drug: pre-operative therapy

INTERVENTIONS:
Drug: pre-operative therapy — pre-operative therapy includes pre-operative chemotherapy, radiation, endocrine therapy, target therapy and other anti-tumor therapy

SUMMARY:
This is a prospective and retrospective study to evaluate the effect of pre-operative therapy on response and survival, and compare the difference in response and survival by pre-operative regimen or by patient's clinicopathological characteristic in early or advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Female, Aged ≥18 years
* Histologically confirmed primary breast cancer
* Plan to receive pre-operative therapy
* Adequate organ function

Exclusion Criteria:

* History of neurological or psychological disease, including epilepsy or dementia
* Not suitable to participate in this study judged by investigators

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be selected from the hospital where they are treated
Sampling Method: Probability Sample
Enrollment: 488 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2030-11 (Estimated); Study Completion 2030-11 (Estimated)

PRIMARY OUTCOMES:
Pathologic Complete Response | at surgery
  ypT0 ypN0, ypT0/is ypN0

SECONDARY OUTCOMES:
Objective response rate | from the start of pre-operative treatment until the completion of surgery up to 6 months
  the rate of complete response and partial response
Disease-free Survival | From surgery until time of event up to 8 years
  Disease-free survival time is defined as the time from date of randomization until the first occurrence of disease recurrence, distant metastasis and death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, School of Medicine, Shanghai Jiaotong University, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chen X, Zhao Y, Wang Y, Ye Y, Xu S, Zhou L, Lin Y, Lu J, Yin W. Serum lipid ratios as novel prognostic biomarkers for patients with locally advanced breast cancer treated with neoadjuvant therapy. Postgrad Med. 2024 Jun;136(5):541-550. doi: 10.1080/00325481.2024.2370235. Epub 2024 Jun 24. PMID 38912905